CLINICAL TRIAL: NCT06797544
Title: The Clinical Effect of Intralesional Injection of Levofloxacin for the Management of Cutaneous Leishmaniasis: Single Arm Open-label Trial
Brief Title: Intralesional Injection of Levofloxacin for the Management of Cutaneous Leishmaniasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hayder Adnan Fawzi (Other)
Responsible Party: Sponsor-Investigator, Hayder Adnan Fawzi, Ass Prof, Al-Mustafa University College
Organization: Al-Mustafa University College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM25-001; apporval no (57) (Other: Research Ethical Approval of Mustansiriyah University/ College of Pharmacy)
Record Dates: First submitted 2025-01-17; First posted 2025-01-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Ofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intralesional levofloxacin (Experimental): Intralesional levofloxacin (5 mg/ml, 100 ml, Tavanic®, Sanofi, France) will be injected into each lesion based on its size (5 mg/cm2). The infiltration of intralesional dose will be given once weekly for up to 6 weeks. Treatment will be stopped in patients cured before 6 weeks of treatment, and patients were only asked to come for lesion assessment. A fine insulin needle will be used to infiltrate the lesion.
  Interventions: Drug: Levofloxacin 0.5%

INTERVENTIONS:
Drug: Levofloxacin 0.5% — Intralesional levofloxacin (5 mg/ml, 100 ml, Tavanic®, Sanofi, France) will be injected into each lesion based on its size (5 mg/cm2). The infiltration of intralesional dose will be given once weekly for up to 6 weeks. Treatment will be stopped in patients cured before 6 weeks of treatment, and patients were only asked to come for lesion assessment. A fine insulin needle will be used to infiltrate the lesion.
  The lesion will be thoroughly infiltrated with the drug solution until the base will be completely blanched. Depending on the lesion size, the amount of solution required ranged from 0.2 to 4.0 ml per lesion. No local anesthesia was added. The solutions were injected intralesionally and not subcutaneously.
  Other Names: Tavanic

SUMMARY:
Aim of the study to evaluate the effectiveness of intralesional levofloxacin 0.5% solution as a local injection in treating cutaneous leishmaniasis.

In an open-label single-arm clinical trial, all patients were given intralesional levofloxacin injections; the patients had cutaneous leishmaniasis lesions. Each lesion was considered a case in the final analysis. Each lesion will be followed up for 90 days (censor endpoint) or until the lesions are cured.

Intralesional levofloxacin (5 mg/ml, 100 ml, Tavanic®, Sanofi, France) will be injected into each lesion based on its size (5 mg/cm2). The infiltration of intralesional dose will be given once weekly for up to 6 weeks. Treatment will be stopped in patients cured before 6 weeks of treatment. A fine insulin needle will be used to infiltrate the lesion.

DETAILED DESCRIPTION:
Local therapies have been recommended by the World Health Organization (WHO), the Pan American Health Organization, and other experts as an alternative to systemic drugs in patients with at least four lesions smaller than 4 cm in diameter, especially when the face or joints are not affected. Usually, they are easy to use and have a lower risk, toxicity, and cost compared to traditional therapies. Local treatment includes thermotherapy, cryotherapy, and topical and intralesional drugs. The last approach is effective and safe in localized forms

ELIGIBILITY:
Inclusion Criteria:

* Patients with single or multiple (less than seven lesions) lesions of cutaneous leishmaniasis and patients ranging in age from 20 to 75 years old.

Exclusion Criteria:

* Patients who received anti-leishmaniasis treatment locally or systemically for the last month before this study and patients on prolonged corticosteroid therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-09 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate | From enrollment to the end of treatment up to 90 days.
  Patients were followed weekly up to 90 days after the first injection; four parameters were used for assessment as follows according to Sharquie modified leishmania score: 1. Measure the size of the lesion through the surface area 2. Measurement of the induration of the lesion 3. Assess the degree of erythema of the lesion 4. Assess the presence and absence of ulceration The obtained data is converted from numbers into scores. The total score was calculated by adding individual scores. Score 13-16: Mild response. Score 9-12: Moderate response. Score 5-8: Marked response. Score 0-4: Complete response & clearance Both marked and complete responses are considered as a cure

CONTACTS AND LOCATIONS:
Locations (1):
- Mustansiriyah University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided